CLINICAL TRIAL: NCT04186000
Title: Open-label Phase 2 Study to Evaluate the Immunogenicity and Safety of a Prophylactic Vaccination of Health Care Providers by Administration of a Heterologous Vaccine Regimen Against Ebola in the Democratic Republic of the Congo
Brief Title: Study to Evaluate the Immunogenicity and Safety of a Heterologous Vaccine Regimen Against Ebola
Acronym: EBOVAC3DRC
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Universiteit Antwerpen (Other)
Collaborators: Johnson & Johnson (Industry); Ace Africa (Other); Innovative Medicines Initiative (Other); Coalition for Epidemic Preparedness Innovations (Other); University of Kinshasa (Other)
Responsible Party: Principal Investigator, Pierre Van Damme, clinical professor, Universiteit Antwerpen
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: VAC52150EBL2007; EDMS-ERI-176345633 (Other: EDMS)
Record Dates: First submitted 2019-12-01; First posted 2019-12-04 (Actual); Last update posted 2023-01-04 (Actual); Status verified 2023-01

CONDITIONS: Ebola Virus Disease
Keywords: Ad26.ZEBOV; MVA-BN-Filo; DRC; health care providers
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Intervention Model Description: All participants receive a heterologous vaccine regimen with Ad26.ZEBOV as first vaccine followed by second dose with MVA-BN-Filo administered 56 days later (Day 57). After randomization (1:1), a booster vaccination with Ad26.ZEBOV will be executed at 1 year post first dose or 2 years post first dose.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- group 1 (Experimental): Booster vaccine with AD26.ZEBOV after 1 year
  Interventions: Biological: Ad26.ZEBOV vaccine
- group 2 (Experimental): Booster vaccine with AD26.ZEBOV after 2 years
  Interventions: Biological: Ad26.ZEBOV vaccine

INTERVENTIONS:
Biological: Ad26.ZEBOV vaccine — The booster vaccination with Ad26.ZEBOV (5x10^10 vp, same dosage as during the first dose) will be given at 1 year after the first dose or 2 years post-first dose.

SUMMARY:
This Phase 2 study aims to improve preparedness for future Ebola outbreaks by vaccination of a well-known population at risk, ie, a cohort of health care providers (HCP) (such as primary, emergency, and community health care workers) who may be exposed to Ebola in the event of a future outbreak in the Democratic Republic of the Congo (DRC). This study will enhance the immunogenicity database by investigating the kinetics of the humoral immune response. The study will contribute to the safety database (serious adverse events) for VAC52150 following a heterologous vaccine regimen with Ad26.ZEBOV as first vaccine followed by second dose with MVA-BN-Filo administered 56 days later (Day 57). Additionally, after randomization (1:1), a booster vaccination with Ad26.ZEBOV will be executed at 1 year post first dose or 2 years post first dose.

DETAILED DESCRIPTION:
This study is an open-label, monocentric (in Tshuapa province, DRC), phase 2 study to evaluate the immunogenicity and safety of Ad26.ZEBOV (5x1010 viral particles [vp]) as first dose and MVA-BN-Filo (1x108 50% infectious units [Inf U]) as second dose vaccination at a 56-day interval in health care providers (HCP) who may be exposed to Ebola in the event of a future Ebola outbreak in DRC. Additionally, after randomization (1:1) a booster of Ad26.ZEBOV (5x1010 vp) will be offered at respectively 1 year or 2 years after the first dose.

A planned total number of approximately 700 participants will be recruited from the Tshuapa province in DRC. At Day 1, interested participants will be assessed for their understanding of the study, will provide consent, their general health will be evaluated by the investigator, medical history (including vaccination history) will be collected, urine pregnancy testing for women of childbearing potential will be performed. Further during this first visit, vital signs will be measured and a blood sample for baseline immunogenicity assessment will be taken for testing of binding antibody level against EBOV GP using FANG ELISA, presence of pre-existing Human anti-EBOV GP IgG and anti-EBOV NP IgG using ELISA and on the first 100 subjects additionally testing for neutralizing antibody level against Ad26 and MVA vectors using respectively Ad26 VNA and MVA PRNT. Subsequently, a blood sample for baseline safety assessment will be performed to test hemoglobin, hematocrit, blood cell count (red and white), platelet count, urea, creatinine and transaminases. After these primary assessments, they will be vaccinated with first dose Ad26.ZEBOV vaccine. They will be given instructions to contact the study team for any serious adverse event that occurs up until 6 months after each vaccination, or in case of pregnancy of the participant during the study. Lastly on day 1, randomization will be performed (1:1) to determine timing of the booster vaccine at 1 year or 2 years after first dose. Contact information will be verified and an appointment for the second dose on Day 57 will be arranged.

At Day 57, participants will return to the study site for urine pregnancy testing for women of childbearing potential, vital signs measurement, assessment of safety (serious adverse events), for a blood sample for immunogenicity assessment (the binding antibody levels against EBOV GP using FANG ELISA) and afterwards administration of the MVA-BN-Filo vaccination, and they will be reminded to contact the study team for any serious adverse event that occurs, or in case of pregnancy of the participant during the study. Contact information will be verified and an appointment for the 21-day post-dose 2 (Day 78) visit will be arranged.

At 21 days post-dose 2 (Day 78), all participants will return to the study site for assessment of safety (serious adverse events) and collection of a blood sample for immunogenicity assessment. Contact information will be re-verified. They will be reminded to contact the study team for any serious adverse event that occurs, or in case of pregnancy of participant.

At approximately 6 months post-dose 2 vaccination, participants will be contacted by phone to inquire about any occurrence of serious adverse events, and to confirm contact information for additional follow up at 1 year post-first dose vaccination. At 1 year after first vaccine dose, a blood sample will be collected for immunogenicity assessment of all participants (where applicable, pre-administration of the booster dose).

Depending on randomization performed at Day 1, the booster vaccination with Ad26.ZEBOV (5x1010 vp) will be given at 1 year after the first dose or 2 years post-first dose. Participants will be asked to collect solicited adverse events in a participant diary starting on the day of vaccination and continuing for the subsequent 7 days. At day 8 post booster (PB) the safety data including solicited adverse events will be reviewed and a blood sample for immunogenicity will be taken to document the immunity response. At 6 months PB, the participants will be contacted by phone and questioned about any serious adverse events that have occurred since the last vaccination. For all participants at 2 years after first dose, a sample will be collected for immunogenicity assessment (where applicable, pre-administration of the booster dose).

The total duration of the study is 2 years and 6 months post-first dose.

ELIGIBILITY:
Inclusion Criteria:

* The participant must pass the Test of Understanding (TOU).
* Each participant must sign an informed consent form (ICF) indicating that he or she understands the purpose of, and procedures required for, the study and is willing to participate in the study. In case the participant cannot read or write, the procedures must be explained and informed consent must be witnessed by a trusted literate third party not involved with the conduct of the study.
* Participant must be a man or woman aged 18 years or older.
* Participant must be a documented health care provider in DRC.
* Participant must be healthy in the investigator's clinical judgment and on the basis of vital signs assessed at day 1 screening.
* Before vaccination, a woman must be either:

Of childbearing potential and practicing (or intending to practice) a highly effective method of birth control consistent with local regulations and/or local culture regarding the use of birth control methods for participants in clinical studies, beginning at least 28 days prior to vaccination and during the study up to at least 3 months after the first (or only) vaccination (Ad26.ZEBOV) and 1 month after the MVA-BN-Filo vaccination (if applicable); and then starting again 14 days before the booster vaccination until 3 months after the booster vaccination.

OR Not of childbearing potential: postmenopausal (amenorrhea for at least 12 months without alternative medical cause); permanently sterilized (eg, bilateral tubal occlusion [which includes tubal ligation procedures as consistent with local regulations], hysterectomy, bilateral salpingectomy, bilateral oophorectomy); OR otherwise be incapable of pregnancy.

* Woman of childbearing potential must have a negative urine β-human chorionic gonadotropin (β-hCG) pregnancy test immediately prior to each study vaccine administration.
* Participant must be available and willing to participate for the duration of the study.
* Participant must be willing and able to comply with the protocol requirements, including the prohibitions and restrictions specified in Section 4.3.
* Participant must be willing to provide verifiable identification.
* Participant must have a means to be contacted.

Exclusion Criteria:

* Known history of Ebola virus disease.
* Having received any experimental candidate Ebola vaccine less than 3 months prior to the screening at the first visit.
* Having received any experimental candidate Ad26-vaccine in the past. Known allergy or history of anaphylaxis or other serious adverse reactions to vaccines or vaccine products (including any of the constituents of the study vaccines [eg, polysorbate 80, ethylenediaminetetraacetic acid (EDTA) or L-histidine for Ad26.ZEBOV vaccine; and tris (hydroxymethyl)-amino methane (THAM) for MVA BN-Filo vaccine]), including known allergy to egg, egg products and aminoglycosides.
* Presence of acute illness (this does not include minor illnesses such as mild diarrhea or mild upper respiratory tract infection) or temperature ≥38.0ºC on Day 1. Participants with such symptoms will be excluded from enrollment at that time, but may be rescheduled for enrollment at a later date if feasible.
* Pregnant or breastfeeding women, or women planning to become pregnant while enrolled in this study until at least 3 months after the Ad26.ZEBOV vaccination or 1 month after MVA-BN-Filo.
* Presence of significant conditions or clinically significant findings at screening or vital signs for which, in the opinion of the investigator, participation would not be in the best interest of the participant (eg, compromise the safety or well-being) or that could prevent, limit, or confound the protocol-specified assessments.
* Major surgery (per the investigator's judgment) within the 4 weeks prior to screening, or planned major surgery during the study (from the start of screening onwards).
* Post-organ and/or stem cell transplant whether or not with chronic immunosuppressive therapy.
* Received an investigational drug or investigational vaccines or used an invasive investigational medical device within 3 months prior to screening, or current or planned participation in another clinical study during the study.
* History of chronic urticaria (recurrent hives).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 699 (Actual)
Dates: Start 2019-12-18 (Actual); Primary Completion 2020-04-25 (Actual); Study Completion 2022-10-12 (Actual)

PRIMARY OUTCOMES:
Binding antibody responses post-dose 2 vaccination with MVA-BN-Filo | 21 days post-dose 2 vaccination
  To assess binding antibody levels against the EBOV GP using FANG ELISA

SECONDARY OUTCOMES:
Safety of a heterologous vaccine regimen utilizing Ad26.ZEBOV as dose 1, MVA-BN-Filo as dose 2 and Ad26.ZEBOV as booster dose 3 | The entire clinical study for SAE reporting and until 7 days post booster for solicited local and system adverse events
  To assess serious adverse events (SAE) during the entire clinical study and to assess solicited local and systemic adverse events until 7 days post booster/dose 3 vaccination with Ad26.ZEBOV
Binding antibody responses after booster vaccination with Ad26.ZEBOV | 7 days post-booster vaccination
  To assess binding antibody levels against the EBOV GP using FANG ELISA

CONTACTS AND LOCATIONS:
Overall Officials: Hypolite Mavoko Muhindo, Dr., Principal Investigator — University of Kinshasa, Tropical Medicine Department
Locations (1):
- Hôpital Général de Référence de Boende, Boende, Province de La Tshuapa, Democratic Republic of the Congo

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Baize S, Pannetier D, Oestereich L, Rieger T, Koivogui L, Magassouba N, Soropogui B, Sow MS, Keita S, De Clerck H, Tiffany A, Dominguez G, Loua M, Traore A, Kolie M, Malano ER, Heleze E, Bocquin A, Mely S, Raoul H, Caro V, Cadar D, Gabriel M, Pahlmann M, Tappe D, Schmidt-Chanasit J, Impouma B, Diallo AK, Formenty P, Van Herp M, Gunther S. Emergence of Zaire Ebola virus disease in Guinea. N Engl J Med. 2014 Oct 9;371(15):1418-25. doi: 10.1056/NEJMoa1404505. Epub 2014 Apr 16. PMID 24738640
- [Result] Baden LR, Walsh SR, Seaman MS, Tucker RP, Krause KH, Patel A, Johnson JA, Kleinjan J, Yanosick KE, Perry J, Zablowsky E, Abbink P, Peter L, Iampietro MJ, Cheung A, Pau MG, Weijtens M, Goudsmit J, Swann E, Wolff M, Loblein H, Dolin R, Barouch DH. First-in-human evaluation of the safety and immunogenicity of a recombinant adenovirus serotype 26 HIV-1 Env vaccine (IPCAVD 001). J Infect Dis. 2013 Jan 15;207(2):240-7. doi: 10.1093/infdis/jis670. Epub 2012 Nov 2. PMID 23125444
- [Result] Friedrich BM, Trefry JC, Biggins JE, Hensley LE, Honko AN, Smith DR, Olinger GG. Potential vaccines and post-exposure treatments for filovirus infections. Viruses. 2012 Sep;4(9):1619-50. doi: 10.3390/v4091619. Epub 2012 Sep 21. PMID 23170176
- [Result] Kohl KS, Walop W, Gidudu J, Ball L, Halperin S, Hammer SJ, Heath P, Varricchio F, Rothstein E, Schuind A, Hennig R; Brighton Collaboration Local Reaction Working Group for Swelling at or near Injection Site. Swelling at or near injection site: case definition and guidelines for collection, analysis and presentation of immunization safety data. Vaccine. 2007 Aug 1;25(31):5858-74. doi: 10.1016/j.vaccine.2007.04.056. Epub 2007 May 11. No abstract available. PMID 17548132
- [Result] Kohl KS, Walop W, Gidudu J, Ball L, Halperin S, Hammer SJ, Heath P, Hennig R, Rothstein E, Schuind A, Varricchio F; Brighton Collaboration Local Reactions Working Group for Induration at or near Injection Site. Induration at or near injection site: case definition and guidelines for collection, analysis, and presentation of immunization safety data. Vaccine. 2007 Aug 1;25(31):5839-57. doi: 10.1016/j.vaccine.2007.04.062. Epub 2007 May 8. No abstract available. PMID 17553602
- [Result] Marcy SM, Kohl KS, Dagan R, Nalin D, Blum M, Jones MC, Hansen J, Labadie J, Lee L, Martin BL, O'Brien K, Rothstein E, Vermeer P; Brighton Collaboration Fever Working Group. Fever as an adverse event following immunization: case definition and guidelines of data collection, analysis, and presentation. Vaccine. 2004 Jan 26;22(5-6):551-6. doi: 10.1016/j.vaccine.2003.09.007. No abstract available. PMID 14741143
- [Result] Stittelaar KJ, Kuiken T, de Swart RL, van Amerongen G, Vos HW, Niesters HG, van Schalkwijk P, van der Kwast T, Wyatt LS, Moss B, Osterhaus AD. Safety of modified vaccinia virus Ankara (MVA) in immune-suppressed macaques. Vaccine. 2001 Jun 14;19(27):3700-9. doi: 10.1016/s0264-410x(01)00075-5. PMID 11395204
- [Result] Verheust C, Goossens M, Pauwels K, Breyer D. Biosafety aspects of modified vaccinia virus Ankara (MVA)-based vectors used for gene therapy or vaccination. Vaccine. 2012 Mar 30;30(16):2623-32. doi: 10.1016/j.vaccine.2012.02.016. Epub 2012 Feb 17. PMID 22342706
- [Result] Hoff NA, Mukadi P, Doshi RH, Bramble MS, Lu K, Gadoth A, Sinai C, Spencer D, Nicholson BP, Williams R, Mossoko M, Ilunga-Kebela B, Wasiswa J, Okitolonda-Wemakoy E, Alfonso VH, Steffen I, Muyembe-Tamfum JJ, Simmons G, Rimoin AW. Serologic Markers for Ebolavirus Among Healthcare Workers in the Democratic Republic of the Congo. J Infect Dis. 2019 Jan 29;219(4):517-525. doi: 10.1093/infdis/jiy499. PMID 30239838
- [Derived] Lariviere Y, Matuvanga TZ, Osang'ir BI, Milolo S, Meta R, Kimbulu P, Robinson C, Katwere M, McLean C, Lemey G, Matangila J, Maketa V, Mitashi P, Van Geertruyden JP, Van Damme P, Muhindo-Mavoko H. Ad26.ZEBOV, MVA-BN-Filo Ebola virus disease vaccine regimen plus Ad26.ZEBOV booster at 1 year versus 2 years in health-care and front-line workers in the Democratic Republic of the Congo: secondary and exploratory outcomes of an open-label, randomised, phase 2 trial. Lancet Infect Dis. 2024 Jul;24(7):746-759. doi: 10.1016/S1473-3099(24)00058-6. Epub 2024 Mar 26. PMID 38552653
- [Derived] Lariviere Y, Matuvanga TZ, Lemey G, Osang'ir BI, Vermeiren PP, Milolo S, Meta R, Kimbulu P, Esanga E, Matangila J, Van Geertruyden JP, Van Damme P, Maketa V, Muhindo-Mavoko H, Mitashi P. Conducting an Ebola vaccine trial in a remote area of the Democratic Republic of the Congo: Challenges, mitigations, and lessons learned. Vaccine. 2023 Dec 12;41(51):7587-7597. doi: 10.1016/j.vaccine.2023.11.030. Epub 2023 Nov 22. PMID 37993355
- [Derived] Zola Matuvanga T, Lariviere Y, Lemey G, De Bie J, Milolo S, Meta R, Esanga E, Vermeiren PP, Thys S, Van Geertruyden JP, Van Damme P, Maketa V, Matangila J, Mitashi P, Muhindo-Mavoko H. Setting-up an Ebola vaccine trial in a remote area of the Democratic Republic of the Congo: Challenges, mitigations, and lessons learned. Vaccine. 2022 May 31;40(25):3470-3480. doi: 10.1016/j.vaccine.2022.04.094. Epub 2022 May 9. PMID 35550847
- [Derived] Lariviere Y, Zola T, Stoppie E, Maketa V, Matangila J, Mitashi P, De Bie J, Muhindo-Mavoko H, Van Geertruyden JP, Van Damme P. Open-label, randomised, clinical trial to evaluate the immunogenicity and safety of a prophylactic vaccination of healthcare providers by administration of a heterologous vaccine regimen against Ebola in the Democratic Republic of the Congo: the study protocol. BMJ Open. 2021 Sep 28;11(9):e046835. doi: 10.1136/bmjopen-2020-046835. PMID 34588237
- [Derived] Zola Matuvanga T, Johnson G, Lariviere Y, Esanga Longomo E, Matangila J, Maketa V, Lapika B, Mitashi P, Mc Kenna P, De Bie J, Van Geertruyden JP, Van Damme P, Muhindo Mavoko H. Use of Iris Scanning for Biometric Recognition of Healthy Adults Participating in an Ebola Vaccine Trial in the Democratic Republic of the Congo: Mixed Methods Study. J Med Internet Res. 2021 Aug 9;23(8):e28573. doi: 10.2196/28573. PMID 34378545
- See also: IMVANEX suspension for injection. UK Summary of Product Characteristics. — https://www.ema.europa.eu/en/documents/product-information/imvanex-epar-product-information_en.pdf
- See also: MVA-BN® (Modified Vaccinia Ankara - Bavarian Nordic). — http://www.bavarian-nordic.com/pipeline/technology/mva-bn.aspx
- See also: WHO Fact Sheet No103 Ebola Virus Disease 2014 — https://www.who.int/en/news-room/fact-sheets/detail/ebola-virus-disease